CLINICAL TRIAL: NCT03485430
Title: Tapering of Prescribed Opioids in Patients With Long-term Non-malignant Pain - Efficacy and Effects on Pain, Pain Cognitions, and Quality of Life (TOPIO): a Study Protocol for a Randomized Controlled Clinical Trial With a 12 Month Follow-up
Brief Title: Tapering From Long-term Opioid Therapy in Chronic Pain Population. Randomized Controlled Trial With 12 Months Follow up
Acronym: TOPIO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Lund University (Other); University Hospital, Linkoeping (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7206093515
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain; Analgesics, Opioid; Opioid Withdrawal; Opioid Use; Substance Use Disorders
MeSH Terms: conditions — Chronic Pain; Substance-Related Disorders | interventions — Drug Tapering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Receives tapering of opioid dose at baseline
  Interventions: Behavioral: Tapering
- Control (No Intervention): Waiting-list. Receives tapering after 4 months.

INTERVENTIONS:
Behavioral: Tapering — Tapering with follow up by nurse at weekly basis in beginning of tapering. Tapering in an outpatient setting. Follow-up to doctor after four months.
  Arms: Intervention

SUMMARY:
This randomized controlled study compares tapering of long-term opioid therapy in a population with chronic non-cancer pain with control group constituted of waiting list. Half of participants receives intervention at baseline and the other half are controls but receives intervention after 4 months. Ethical approval to follow up excluded participants denying tapering at baseline.

DETAILED DESCRIPTION:
Chronic non-cancer pain is a major problem in society and a common cause to seek health care. The suffering is complex as it, besides pain, often includes psychological symptoms and may decrease the ability to participate in work life. Pharmacological treatments have limited possibilities to ease suffering. Opioids used in this population have evidence to ease pain and to some extent increase physical ability when used in limited treatment periods and in selected patients. Medium to long-term opioid therapy, extended beyond three months, lack evidence of easing pain or increase physical ability.

The current study is conducted on three specialized pain care units (Skane University Hospital; Lund, Sahlgrenska University Hospital Gothenburg and University Hospital, Linkoeping) and aims at taper long-term opioid therapy with support from physician and nurse and study the effects of tapering.

Method: Randomized controlled study, without concealment. Waiting-list constitutes the control-group. Intervention means tapering with a motivated patient. Follow up at four and twelve months.

Primary end-point: collected opioid prescriptions registered in The National Board of Health and Welfare registry expressed in milligram of morphine equivalent.

Secondary end-point: Data will be retrieved from the Swedish Quality Registry for Pain Rehabilitation. The database contains participants' self-report of variables measuring the impact of rehabilitation on depressive symptoms, anxiety, rating of pain and acceptance to pain. Assessments are made prior to, at the end of and one year after discharge of the rehabilitation program.

As denying tapering or participation is shown to be as common as decision to taper drugs at baseline an extended ethical approval was acquired also retrospective. This approval covers obtaining collected prescribed medication and prescribed opioid replacement therapy (Buprenorphine or Methadone) after one year. The study may describe the excluded population better this way.

ELIGIBILITY:
Inclusion Criteria:

A long-term opioid therapy with daily intake due to chronic pain condition, by prescription. Willing to enter an intervention aiming at taper opioid therapy.

Exclusion Criteria:

No daily intake of opioids. Shorter duration of opioid therapy than 3 months. Repeated intake of non-prescribed opioids or other illegal drugs. Refusal to perform drug-screening Perceived medical risks of waiting with tapering of opioids (e.g: raising opioid doses after acute pancreatitis caused by excessive alcohol intake or kidney disease stage 4-5 in combination with excessive alcohol intake and high doses of opioids).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 12 months
  Data retrieved from National Boars of Health and Welfare, collected prescribed opioid drugs
Opioid consumption | 4 months
  Self reported consumption

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 12 months
  NPRS was used to capture the patient's level of pain intensity. Patients rate their average level of pain the last week. The 11-point scale spans from the left with the phrase "no pain" i.e. 0 and on the right to the phrase "worst imaginable pain" i.e. 10.

OTHER OUTCOMES:
Hospital Anxiety and Depression scale (HADS) | 12 months
  HADS was constructed for patients in medical settings. It entails 14-item measures of anxiety (7 items) and depression (7 items) symptoms over the course of a week. Items are rated on a four-point scale (0 = not all; 3 = very often) and the anxiety and depression subscales range from 0 to 21. Higher scores indicate greater severity.
Tampa Scale for Kinesiophobia (TSK) | 12 months
  The TSK employs a 4-point Likert scale, with scoring options ranging from 1 (strongly disagree) to 4 (strongly agree) and encompasses 17 items related to pain, fear of movement and re-injury. The total score of the original 17-item version ranges between 17 and 68, with a higher score indicating a higher degree of Kinesiophobia.
Pain Catastrophizing Scale (PCS) | 12 months
  The PCS comprises 13 items that are rated from 0 to 4 with the endpoints 0 ("Never") to 4 ("All the time") and was constructed to assess pain-related catastrophizing (48). Catastrophizing include three factors: (a) Helplessness i.e. perceived helplessness in situations when pain is present (six items); (b) Rumination, concerning vigilance toward the pain experience (four items) ; and (c) Magnification i.e. the tendency to magnify the threat value of pain (three items). The total score ranges from 0-52 points with a higher score indicating a higher degree of catastrophizing.
Chronic Pain Acceptance Questionnaire (CPAQ-8) | 12 months
  Pain acceptance measures two main classes of behaviors represented by respective subscales: Activity Engagement (score range: 0-24), and Pain Willingness (inverted score range: 0-24). The items are rated from 0 (never true) to 6 (always true) and higher values indicate higher acceptance to chronic pain.
Perceptions of health | 12 months
  RAND-36 is a modern translation of SF-36. RAND-36 encompasses questions from eight domains (subscales) i.e. physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE) and mental health (MH). The scores are subsequently transformed in a standardized way into a 0-100 scale where higher scores indicate better health.

CONTACTS AND LOCATIONS:
Overall Officials: Åsa IRingqvist, MD, PhD, Study Chair — Lund University
Locations (3):
- Sweden (3):
  - Lund University Hospital, Lund, Skåne County
  - Paincentre Sahlgrenska University Hospital, Gothenburg, Västra Götaland County
  - Pain and rehabilitation centre Linköping University Hospital, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henrik G, Patrik M, Anders H, Ulf J, Marcelo RF, Asa R. Tapering of prescribed opioids in patients with long-term non-malignant pain (TOPIO)-efficacy and effects on pain, pain cognitions, and quality of life: a study protocol for a randomized controlled clinical trial with a 12-month follow-up. Trials. 2021 Jul 28;22(1):503. doi: 10.1186/s13063-021-05449-5. PMID 34321058